CLINICAL TRIAL: NCT00013741
Title: The MI-HEART Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Library of Medicine (NLM) (NIH)
Allocation: Randomized | Masking: Double
Other Study IDs: 9511; N01-LM-93534
Record Dates: First submitted 2001-03-28; First posted 2001-03-30 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2003-02

CONDITIONS: Myocardial Infarction; Coronary Disease
Keywords: Acute Myocardial Infarction; Diabetes Mellitus; Renal Dialysis; Heart Attack; Coronary Heart Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Diabetes Mellitus

INTERVENTIONS:
Behavioral: Tailored Education Messages

SUMMARY:
The purpose of the study is to examine ways in which a clinical information system can help patients better recognize the signs and symptoms of an acute myocardial infarction (heart attack) and to take actions to decrease morbidity and mortality that may be related to delay in seeking treatment. The software-based intervention will use the best scientific evidence to create tailored strategies using a patient's specific health data. This approach is based on well-established cognitive and behavioral educational models.

ELIGIBILITY:
Inclusion Criteria

* Patients at high-risk for an acute myocardial infarction, including any 2 of these risk factors: males age > 45; females age >55; family history of premature coronary heart disease (CHD); current cigarette smoker; hypertension; or elevated total cholesterol with low HDL and/or high LDL.

OR have:

* Active angina (chest pain due to coronary heart disease)
* History of coronary heart disease according to the treating physician
* Past history of myocardial infarction documented by electrocardiogram or arteriography
* Diabetes Mellitus
* Renal dialysis

Exclusion Criteria

* Hospitalization within previous 4 weeks
* Persons living in a home with previously enrolled patients
* Patients disoriented to person, place, or time at onset of study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55

CONTACTS AND LOCATIONS:
Overall Officials: James J. Cimino, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, Department of Medical Informatics, New York, New York, United States